CLINICAL TRIAL: NCT03035747
Title: Russian Registry of Treatment of Chronic Venous Diseases
Brief Title: Ongoing Registry of Treatment of Chronic Venous Diseases
Acronym: RRT CVD
Status: Recruiting | Type: Observational
Sponsor: Medalp Private Surgery Clinic (Other)
Collaborators: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Evgeny Ilyukhin, Сhief surgeon Medalp Private Surgery Clinic, Medalp Private Surgery Clinic
Other Study IDs: A001
Record Dates: First submitted 2017-01-25; First posted 2017-01-30 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Varicose Veins of Lower Limb
Keywords: registry; varicose veins; conventional surgery; thermal ablation; radiofrequency; laser; sclerotherapy
MeSH Terms: conditions — Varicose Veins | interventions — Sclerotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: conventional surgery — high ligation and stripping of incompetent saphenous veins
Procedure: endovenous laser ablation — endovenous laser ablation of incompetent saphenous veins
Procedure: sclerotherapy — ultrasound guided or catheter or or any other methods sclerotherapy of incompetent saphenous or varicose veins
Procedure: endovenous radiofrequency ablation — endovenous radiofrequency ablation of incompetent saphenous veins
Procedure: phlebectomy — hooks phlebectomy of varicose veins

SUMMARY:
Ongoing registration of patients with varicose veins disease treated by means of conventional surgery, endovenous thermal ablations, sclerotherapy, non-tumescent non-thermal methods

DETAILED DESCRIPTION:
Data of patients treated in different Russian medical centers are entered in a prospective digital database, and continuously updated.

There is planned to conduct prospective randomized, cohort and observational studies on the site of register

ELIGIBILITY:
Inclusion Criteria:

* Varicose veins with any source of pathological reflux, C2 - C6 according to the CEAP classification

Exclusion Criteria:

* no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing interventions in cases varicose vein disease
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2036-07 (Estimated); Study Completion 2036-07 (Estimated)

PRIMARY OUTCOMES:
Change in patency target veins assessed by duplex ultrasonography in different follow up periods after conventional surgery, endovenous thermal ablations, sclerotherapy or non-tumescent non-thermal methods | Baseline, 3 - 6, 12 months post-intervention

SECONDARY OUTCOMES:
Change in Quality of Life (QoL), assessed by Short form (SF)-36 health survey (optional) | Baseline, 3 and 12 months post-intervention
  The SF-36 is a generic QoL questionnaire.
Change in Venous Clinical Severity Score (VCSS) (optional) | Baseline, 3 and 12 months post-intervention
  The VCSS is a validated scoring system for assessing signs, symptoms and complaints of venous disease.
Change in Quality of Life (QoL), assessed by Aberdeen Varicose Vein Questionnaire (AVVQ) (optional) | Baseline, 3 and 12 months post-intervention
  The AVVQ is a disease-specific QoL questionnaire aimed at venous disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Medalp private surgery clinic, Saint Petersburg, Russia

REFERENCES:
- See also: Russian Register of Treatment of Chronic Venous Diseases (RRT CVD) — http://www.venousregistry.org/
- See also: Russian Phlebological Association (RPA) — https://phlebounion.ru/en/
- See also: Confirmation page about membership of RPA in the International Union of Phlebology — https://www.uip-phlebology.org/society?code=EU